CLINICAL TRIAL: NCT02825589
Title: Effect of Bioelectrical Impedance Analysis-Guided Comparing With Standard Clinical-Guided Dry Weight Assessment on Sleep Quality in Chronic Hemodialysis Patients
Brief Title: BIA-Guided Dry Weight Assessment on Sleep Quality in Chronic Hemodialysis Patients
Acronym: BEDTIME
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ID05-59-12
Record Dates: First submitted 2016-07-03; First posted 2016-07-07 (Estimated); Last update posted 2019-03-08 (Actual); Status verified 2019-03

CONDITIONS: Renal Failure Chronic Requiring Hemodialysis; Poor Quality Sleep
Keywords: BIA; chronic hemodialysis; sleep quality
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- BIA-guided (Experimental): Assessment of target dry weight guided by using bioelectrical impedance analysis (BIA).
  Interventions: Device: BIA
- Standard clinical guided (No Intervention): Assessment of target dry weight guided by clinical evaluation eg. jugular venous pressure, blood pressure, edema etc.

INTERVENTIONS:
Device: BIA — BIA or bioelectrical impedance analysis using electric current through body tissues to estimate body composition particularly body fat and total body water calculating to target body weight.
  Arms: BIA-guided

SUMMARY:
Based on many previous data proving hypervolemia in chronic hemodialysis patients could lead to sleep apnea and poor sleep quality. The investigators conduct this trial to evaluate whether more accurate dry weight assessment with BIA in these patients can lead to better sleep quality (measured by sleep actigraphy and questionnaires). The investigators will enroll 30 chronic hemodialysis patients in hemodialysis unit of Ramathibodi hospital whose age > 18 years with subclinical hypervolemic status and baseline Pittsburgh sleep quality index (PSQI) score > 5 into study. Patients with bed-ridden status, alteration of consciousness and unstable hemodynamics will be excluded. Then eligible patients will be randomized into 2 groups, BIA-guided and standard clinical guided dry weight assessment. The investigators will assess participants' dry weight at beginning of study, 3rd month and 6th month. Sleep actigraphy parameters (eg. total sleep time, sleep efficiency), sleep questionnaires score, left ventricular mass index by echocardiography, ambulatory blood pressure monitoring and blood chemistry results were collected at beginning of study, the end of 1st, 3rd and 6th month. The primary outcome is change of sleep actigraphy parameters between the groups. The secondary outcomes are change of sleep questionnaires scores, change of left ventricular mass index, change of ambulatory BP monitoring and also cardiovascular complications between groups.

DETAILED DESCRIPTION:
This randomized control trial aim to detect the better volume control guided by bioimpedance may improve ambulatory blood pressure control, sleep quality and left ventricular hypertrophy.

ELIGIBILITY:
Inclusion Criteria:

* regular hemodialysis 3 times/week
* PSQI score >5
* Subclinical hypervolemia

Exclusion Criteria:

* bed ridden status
* alteration of consciousness
* unstable hemodynamics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2017-01 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Change of sleep actigraphy parameters | 6 months
  total sleep time, sleep efficiency, fragmentation index

SECONDARY OUTCOMES:
Change of PSQI scores | 6 months
  PSQI or Pittsburgh sleep Quality Index is an instrument for assessment subjective sleep quality in various group of patients.
Change of left ventricular mass index by echocardiography | 6 months
Change of ambulatory blood pressure monitoring | 6 months
Cardiovascular complications | 6 months
  complications which can occur from overestimate of ultrafiltration eg. intradialytic hypotension, arrhythmia, cerebral vascular events, myocardial ischemic events etc.

CONTACTS AND LOCATIONS:
Overall Officials: Arkom Nongnuch, MD, Principal Investigator — Ramathibodi Hospital
Locations (1):
- Ramathibodi hospital, Mahidol university, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sethakarun S, Bijaphala S, Kitiyakara C, Boongird S, Phanachet P, Reutrakul S, Pirojsakul K, Nongnuch A. Effect of bioelectrical impedance analysis-guided dry weight adjustment, in comparison to standard clinical-guided, on the sleep quality of chronic haemodialysis patients (BEDTIME study): a randomised controlled trial. BMC Nephrol. 2019 Sep 2;20(1):211. doi: 10.1186/s12882-019-1405-z. PMID 31474223